CLINICAL TRIAL: NCT00487357
Title: MATCh Parents' Supplemental Survey: Predictors of Smoking in Mexican American Youth
Brief Title: MATCh Parents' Supplemental Survey
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0294
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2012-06

CONDITIONS: Epidemiology
Keywords: Epidemiology; Cancer Prevention; Questionnaire; MATCh; Survey
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MATCh Parents' Supplemental Survey: Parent/Guardian Survey
  Interventions: Behavioral: Supplemental Survey

INTERVENTIONS:
Behavioral: Supplemental Survey — Questionnaire give during home visit to collect behavioral, risk factors and other smoking status data on MATCh parents/guardians.
  Other Names: Questionnaire

SUMMARY:
Primary Objectives:

1. To collect data on health behaviors in the parents of MATCh study participants
2. To collect and/or update risk factor data from the parents of the MATCh study participants.

DETAILED DESCRIPTION:
This research project is for the parents of study participants in the "Predictors of Smoking in Mexican American Youth," also known as the MATCh study.

This research project has three objectives.

These include:

1. collecting data on your health behaviors. Researchers are interested in this information because your health behaviors may influence your children's health behavior;
2. learning about the types of interventions that would be of most use and interest to you and your family; and
3. learning about the most convenient and useful way in which these interventions would be delivered.

Researchers are interested in knowing about the types of interventions that would benefit you and your family because they would like to design future intervention studies that meet your needs and the needs others in your community.

ELIGIBILITY:
Inclusion Criteria:

1. The parent or legal guardian of the child participating in UT MDACC Protocol 2004-0616. Parents/legal guardians will be identified and enrolled after their child is enrolled in protocol 2004-0616.
2. Participants who speak English, Spanish or are bilingual are eligible to participate.

Exclusion Criteria: None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents/guardians of participants in the MATCh study (accompany UT MDACC Protocol 2004-0616, "Predictors of Smoking in Mexican American Youth," also known as the MATCh study).
Sampling Method: Probability Sample
Enrollment: 1215 (Actual)
Dates: Start 2006-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Data collection on health behaviors in the parents of MATCh study participants. | 4 Years

SECONDARY OUTCOMES:
Data collection and/or update risk factors from the parents of the MATCh study participants. | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Sara Strom, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org